CLINICAL TRIAL: NCT03979144
Title: Usability Study of a Self-test Prototype for Human Immunodeficiency Virus (HIV) Screening
Status: Completed | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 003/2017
Record Dates: First submitted 2019-05-20; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Mass Screening
Keywords: Usability; HIV self-test; Prototype
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observational study — This was an observational study of a medical device, through the usability assessment, for the registration of a self-test for the immunodeficiency virus (HIV) screening.

SUMMARY:
It concerns a study to evaluate the usability of an HIV self-test prototype developed from TR DPP® HIV - 1/2 Oral Fluid. The study followed the recommendations of Technical Note No. 20/2016 / GEVIT / GGTPS / ANVISA.

DETAILED DESCRIPTION:
It concerns a study with a mixed method approach to evaluate the usability of a prototype of HIV self-test among lay users. Data collection techniques were performed through observation through videos of lay users conducting self-testing without supervision, a qualitative checklist by participant observation, pre-test and post-test interviews, and closure form. There was no randomization in this study.

The study was conducted by four clinical research sites, distributed in four different states of Brazil in other to obtain a geographic representation: Unidade de Ensaios Clínicos para Imunobiológicos (UECI) at Rio de Janeiro; Centro de Ciências da Saúde da Universidade Federal da Paraíba (UFPB) at Paraíba, Faculdade de Medicina de Botucatu (UNESP) at São Paulo and Centro de Ciências Biológicas e da Saúde da Universidade Estadual do Pará (UEPA) at Pará.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥ 18 years, of both sexes, who agree to participate in the study, after reading, understanding and signing the ICF;
* Individuals who authorized filming during the test.

Exclusion Criteria:

* Illiterates;
* Participants who have already performed any other HIV self-test;
* Health professionals with complete higher education;
* Colorblind individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lay people, that is, individuals without formal technical or scientific training, with different degrees of education, genres and age groups. The user profile included information about the academic / professional training and city / state, of both sexes, selected from characteristics distributed in 4 different groups, including regional variations:
  Group 1: participants with a grade of schooling up to elementary school, in the age group of 18 to 29 years; Group 2: participants with a high school education level, between the ages of 18 and 29; Group 3: participants with educational level up to elementary school, in the age group from 30 years; Group 4: participants with a high school education, in the age group from 30 years of age
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Compliance with self-test execution | Day 1
  Percentage of participants who followed all the steps correctly
Compliance with results interpretation | Day 1
  Percentage of participants who misinterpreted the test result
Compliance with self-test result | Day 1
  Percentage of positive results interpreted as negative
Compliance with self-test steps | Day 1
  Percentage of participants who made mistakes in each of the steps

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana J Fernandes, DSD, MSc, Principal Investigator — Assessoria Clinica / Bio-Manguinhos / Fiocruz
Locations (1):
- Assessoria Clinica / Bio-Manguinhos / Fiocruz, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No